CLINICAL TRIAL: NCT06202274
Title: Clinical Study to Evaluate the Safety and Efficacy of Candela Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PM23001
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hair Reduction; Tattoo Removal; Wrinkle; Acne; Scars; Benign Cutaneous Vascular Lesions; Skin Conditions
MeSH Terms: conditions — Acne Vulgaris; Cicatrix; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment will be performed with commercial products manufactured by Candela and may also include non-Candela products. All devices will be used per the manufacturer's instructions.
  Interventions: Device: Nordlys, Gentle, Picoway, Vbeam, Profound, Profound Matrix, eTwo, Exceed, CO2RE

INTERVENTIONS:
Device: Nordlys, Gentle, Picoway, Vbeam, Profound, Profound Matrix, eTwo, Exceed, CO2RE — Subjects will receive up to twelve (12) treatments at minimum treatment interval of 2 weeks and maximum treatment interval of 12 weeks.

SUMMARY:
This is a non-randomized, multi-center, open-label, prospective clinical study evaluating the clinical treatment with Candela Medical Technology.

DETAILED DESCRIPTION:
Subjects may receive treatment with one applicator or combination of any of the devices and applicators and/or additional commercial devices, products, and procedures. Evaluations may include combination treatments, sequential treatments, split face treatments, exploration of treatment and system parameters, and evaluation of exploratory indications. Treatments may include evaluation of commercial Candela systems with modification in hardware or software and/or treatment outside of treatment guidelines and exploratory indications (off-label) for evaluation of clinical feedback, device components, and treatment outcomes.

Subjects may receive up to twelve (12) treatments. Treatments may occur with a minimum treatment interval of 2 weeks and maximum treatment interval of 12 weeks. The number and interval of treatments will depend upon the device(s), treatment area, and indication to be treated. Follow-up visits may be required per PI discretion. Follow-up visits may occur virtually or in person.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Fitzpatrick skin type I-VI
3. Willingness to provide signed, informed consent to participate in the study
4. Able and willing to comply with the treatment/follow-up schedule and requirements and pre and post treatment instructions.
5. Willing to receive clinical treatments with the study device to be utilized and comply with all study (protocol) requirements.
6. Willingness to allow photographs and/or video of treated areas, and to release their use for scientific/educational and/or promotional/marketing purposes
7. Willing to abstain from any other procedures, medications or topicals in the study treatment areas for the duration of the study which the investigator deems would interfere with the study.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, or breast feeding during the study
2. Skin cancer in the treatment area or history of melanoma in the treatment area
3. History of current cancer and subject has undergone chemotherapy within the last 12 months
4. Severe concurrent conditions, such as cardiac disorders, per investigator discretion
5. Impaired immune system or use of immunosuppressive medications as deemed inappropriate per investigator discretion
6. Herpes Simplex Virus (HSV) in the intended treatment area unless treated following a prophylactic regimen
7. Pacemaker or internal defibrillator or any active electrical implant anywhere in the body if to be treated with an RF based device
8. Superficial metal or other implants in the treatment area, except superficial dental implants, unless these implants can be removed or covered with rolled gauze during treatment if to be treated with an RF based device
9. Active skin condition in the treatment area such as skin infection, sores, psoriasis, eczema, rash, or open wounds as per discretion of the investigator
10. History of abnormal wound healing, keloid, or hypertrophic scar formation, as well as very thin or fragile skin as per discretion of the investigator
11. History of collagen vascular disease or vasculitic disorders as per discretion of the investigator
12. Known allergy to medication to be used during treatments such as allergy to topical anesthetic (e.g. lidocaine)
13. History of systemic corticosteroid therapy in past six months as per discretion of the investigator
14. Tattoos or permanent makeup in the intended treatment area unless to be treated for tattoos or permanent makeup
15. If to be treated for efficacy assessments, history of aesthetics treatments/procedures (e.g. facial resurfacing and deep chemical peeling) within the last 4 months within the intended treatment area, neuromodulator injections (e.g. Botox®), collagen, non-permanent dermal filler, or fat injections or other methods of augmentation with injected bio-material in the treated area within the last 3 months, permanent synthetic fillers (e.g. silicone) in the treatment area, absorbable facial threads within the last 1 year or non-absorbable facial threads within the intended treatment area, or surgery within the intended treatment area. History of prior treatments and procedures will be assessed per investigator discretion.
16. In the opinion of the investigator, the subject is unwilling or unable to adhere to the study requirements or is otherwise unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2028-10-04 (Estimated); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | From the first treatment to the last treatment, up 132 weeks.
  Subject assessment of treatment discomfort/pain immediately post-treatment via Numerical Rating Scale (NRS). Subjects will be presented a horizontal line scale and asked to make a mark along the scale. Subjects will be asked to rate pain from 0 to 10, with 0 equaling no pain and 10 equaling the worst possible pain. A number is obtained by measuring up to the point the participant has indicated.
Post-treatment Assessment Severity Scale | From the first treatment to the last treatment, up to 132 weeks.
  Skin responses including edema, erythema, pinpoint bleeding, purpura/ecchymosis, petechiae, and microscopic epithelial necrotic debris (MENDs) will be assessed immediately after treatment with a post-treatment assessment severity scale: grade 1 means absent, grade 2 means mild, grade 3 means moderate, and grade 3 means severe.

CONTACTS AND LOCATIONS:
Overall Officials: Konika P Schallen, MD, Principal Investigator — Candela Institue for Exellence
Locations (3):
- United States (2):
  - Center for Morden Aesthetic Medicine, Jacksonville, Florida
  - Candela Institue for Excellence, Marlborough, Massachusetts
- Yokneam Candela Clinic, Yokneam Illit, Israel